CLINICAL TRIAL: NCT06079840
Title: Mindfulness Based Stress Reduction App for African American Caregivers
Brief Title: Mindfulness Based Stress Reduction App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: COG Analytics (Other)
Collaborators: Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2R44AG071168-02 (NIH)
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Stress Reduction
Keywords: Digital intervention; Mindfulness; Stress reduction

STUDY DESIGN:
Intervention Model Description: The evaluation will involve a two-group RCT in which 100 African American informal caregivers of PLWHA, who previously participated in a caregiver study will be randomly assigned to one of two conditions: (1) MBSR-AAC app (n=50): Participants will receive the MBSR-AAC app for 8-weeks; or (2) Comparison (n=50): Participants will receive information regarding caregiver services and resources for 8-weeks. Assessments will be conducted with all participants at baseline and 4-, 8-, and 12-weeks post-baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR-AAC app (Experimental): Participants will receive the MBSR-AAC app for 8-weeks.
  Interventions: Device: mindfulness-based stress reduction app
- Comparison (Active Comparator): Participants will receive information regarding caregiver services and resources for 8-weeks.
  Interventions: Device: mindfulness-based stress reduction app

INTERVENTIONS:
Device: mindfulness-based stress reduction app — mobile application (app) for caregivers

SUMMARY:
African American caregivers of people living with HIV/AIDS (PLWHA) have unique needs because they are more likely to experience stressors related to intersecting sources of stigma, discrimination, and caregiving burdens specifically associated with caregiving for PLWHA. The proposed project will enhance and finalize Phase I app development and evaluate its effectiveness in a randomized controlled trial. The project has high public health significance because of its potential to provide an accessible, easy to use mindfulness-based support tool for African American caregivers that could reduce stress, mitigate the harm of intersecting stigmas, and strengthen the caregiver-care recipient relationship.

DETAILED DESCRIPTION:
Building upon prior research regarding mindfulness-based stress reduction interventions, during Phase I, we successfully developed a prototype mobile application (app) for caregivers entitled Mindfulness Based Stress Reduction for African American Caregivers (MBSR-AAC). Based on the Health Stigma and Discrimination Framework, components of the app focus on decreasing stress associated with intersecting sources of stigma, discrimination, and caregiving burdens specifically associated with caregiving for people living with HIV/AIDS (PLWHA). In the present Phase II SBIR study, we will build on Phase I findings to incorporate research-driven enhancements to the app, conduct a feasibility trial of the enhanced app, and conduct a randomized clinical trial to examine the effectiveness of the app in reducing caregiver stress. If proven to be effective, the MBSR-AAC app could have a positive impact on the well-being of African American caregivers that serve as a critical pillar of support for many PLWHA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* African American
* Currently a main unpaid caregiver (defined as providing emotional, physical, and financial support) to a person living with HIV/AIDS.

Exclusion Criteria:

• Inability to provide informed consent (e.g., compromised comprehension).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Perceived caregiver stress | Up to 12 weeks
  The degree to which stressful situations occurred during a specific period of time.
Caregiver self-compassion | Up to 12 weeks
  Caregiver self-kindness, common humanity, mindfulness, self-judgment, isolation, and over-identification during a specific period of time.
Caregiver-care recipient relationships | Up to 12 weeks
  The degree to which the caregiver feels close to the care recipient
Caregiver burden | Up to 12 weeks
  An assessment of various dimensions of caregiver burden (e.g., isolation, relationship strain, privacy, social life, and health).
Caregiver depressive and anxiety symptoms | Up to 12 weeks
  An assessment of caregiver clinical symptoms of depression and anxiety.

SECONDARY OUTCOMES:
Stigma and discrimination | Up to 12 weeks
  An assessment of caregiver general feelings of shame, rejection, and avoidance and an assessment of discrimination experiences in the day-to-day lives of caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Steven B Carswell, Ph.D., Principal Investigator — COG Analytics
Locations (1):
- Friends Research Institute, Baltimore, Maryland, United States